CLINICAL TRIAL: NCT03895632
Title: A Data Collection and Analysis Pilot Study to Indicate Preliminary Characterisation of the Electromyogram Signal in Relation to Needle Position With Respect to the Extraocular Muscles, as Observed During Electromyogram Needle Guided Treatment of Strabismus in Adults
Brief Title: Eye Muscle Needle Electromyogram (EMu) Study
Acronym: EMu
Status: Completed | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 5686
Record Dates: First submitted 2019-01-16; First posted 2019-03-29 (Actual); Results first posted 2020-08-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2019-01

CONDITIONS: Strabismus
Keywords: Extraocular muscle; Electromyogram; Monopolar; Needle guidance; Botulinum toxin; Strabismus
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In some cases, strabismus, or squint, is treated with injections of Botulinum toxin (BTX) to temporarily relax the eye muscle responsible for causing the eye to be pulled to one side. Due to the deep location of the muscles, electromyogram (EMG) needle guidance is used to help ensure the toxin is delivered accurately. EMG needle guidance involves listening to the EMG signal from the tip of the delivery needle - when the needle is in the right place a sound akin to "rain on a tin roof" is heard and the BTX can be injected.

From previous research, clearly clinicians want to improve the technology of this procedure and increase the treatment efficacy and repeatability. After all, the current procedure is imprecise and subjective for what is a small target, with the eye muscles being around 2.5 mm to 4.7 mm in diameter. There may also be an increase in the likelihood of side effects such as droopy eyelids when the toxin spreads beyond the target muscle.

There is a strong need for new knowledge to improve EMG needle guidance in this context. It is hypothesised that the EMG signal could be cleaned and mined for information in real time during the procedure, thus providing the clinician with better information to guide the positioning of the needle before injecting. This pilot study will deliver the knowledge essential to indicate the feasibility of doing this. If feasible, this study will inform a full study with the aim of benefitting patients by allowing new technology to be developed to improve the treatment of strabismus with BTX.

ELIGIBILITY:
Inclusion Criteria:

i. Adults undergoing planned, routine EMG needle guided BTX injection into either lateral or medial rectus muscle for the treatment of strabismus.

ii. Patients being treated by Mr Yagan.

Exclusion Criteria:

- Patients with Chronic progressive external ophthalmoplegia (CPEO) are excluded; a highly attenuated EMG signal is expected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with strabismus being treated with injections of Botulinum toxin.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tristan G Payne, PhD, Principal Investigator — Liverpool University Hospitals NHS Foundation Trust
Locations (1):
- Manchester Royal Eye Hospital, Manchester, United Kingdom

REFERENCES:
- [Background] Pinheiro, J. & Bates, D. (2000) Mixed-Effects Models in S and S-PLUS. Statistics and Computing. New York, NY, USA: Springer-Verlag

RESULTS

PARTICIPANT FLOW:
Groups:
- Observation: Patients with strabismus being treated with injections of Botulinum toxin (BTX).
  BTX dosage varied from 0.5 to 6.0 Units given in a single injection of fluid.
Period: Overall Study
Arm/Group | Observation
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Observation: Participants who were recruited and had their data recorded for this observational study.
Arm/Group | Observation
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 55 [18 to 75]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Sex/Gender data were not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Rectus muscle [Count of Participants; unit: Participants] — Whether the target muscle was the medial rectus or lateral rectus
  Participants
    Medial rectus | 8
    Lateral rectus | 17
Electrode distance [Mean (Full Range); unit: mm] — The measured distance from the participant's outer canthus to the nearest point of the reference electrode
  mm | 13 [10 to 17]

OUTCOME MEASURES:

1. Primary Outcome: α (Slope) Parameter of the Electromyogram (EMG) Signal Power Spectral Density (PSD) Plot as Needle Approaches Then Enters Muscle.
Description: The continuous change in the EMG signal as the needle is (a) distal to, (b) approaches, and (c) enters, the target extraocular muscle.
  Welch's periodogram estimator (Hamming window, 256-point FFT, 50% overlap) was applied to each of the three signal segments described above to obtain an estimate of the PSD of the signal. A robust linear model was fit to estimate the α (slope) parameter of each PSD plot.
Time Frame: Approximately 5 minutes, i.e. immediately prior to needle insertion until Botulinum toxin (BTX) delivery and needle withdrawal
Measure: Number (95% Confidence Interval); unit: log (mV^2 / Hz) / log (Hz)
Arm/Group | Observation
Number analyzed (Participants) | 25
log (mV^2 / Hz) / log (Hz)
  Off-target | 1.49 [1.22 to 1.76]
  Approaching-target | 2.86 [2.59 to 3.13]
  On-target | 3.56 [3.29 to 3.83]
Statistical Analysis 1: Comparison: Observation; The null hypothesis was that α (the slope of the Power Spectral Density (PSD) plot) is not related to signal segment (off-, approaching- and on-target); Test type: Other — A linear mixed-effects model was fit to assess the association between α (the slope of the Power Spectral Density (PSD) plot) and signal segment; p < 0.0001, Linear mixed-effects model — p-value obtained form the Wald statistics of the linear mixed-effects model. The threshold for statistical signifiance was p=0.01

2. Secondary Outcome: Clinical Score of EMG Change
Description: Clinician's score of the step change from baseline EMG to 'active' EMG level heard immediately prior to delivery of Botulinum toxin (BTX) from 1-5. Value from 1 = no significant step change heard, to 5 = a very clear step change heard.
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Observation
Number analyzed (Participants) | 25
score on a scale | 4.6 [3 to 5]

3. Secondary Outcome: Clinical Score of Needle Placement Accuracy
Description: Clinician's score of their confidence in accurate needle placement with respect to the target muscle. Given as a percentage, a higher score indicates more confidence in accurate needle placement.
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: percentage of confidence
Arm/Group | Observation
Number analyzed (Participants) | 25
percentage of confidence | 87.6 [50 to 95]

4. Secondary Outcome: Clinical Score of EMG Quality.
Description: Clinician's score of overall quality of the EMG signal heard during the procedure. A higher score indicates better quality of EMG signal, and is quantified as 1 to 5, where: 1 indicates signal not present and 5 indicates excellent quality EMG signal.
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Observation
Number analyzed (Participants) | 25
score on a scale | 4.5 [3 to 5]

5. Secondary Outcome: Post-treatment Angle of Deviation
Description: Change in participant's angle of deviation following treatment, measured in prism dioptres.
Time Frame: 2 weeks
Population: Data was not collected; it was determined before recruitment began that the value of this data did not merit the significant inconvenience to participants of returning for follow-up measurements.
Arm/Group | Observation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The duration of the Botulinum toxin injection procedure, typically around 5 minutes for each participant.
Arm/Group | Observation
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT03895632/Prot_SAP_000.pdf